CLINICAL TRIAL: NCT06836050
Title: The Effect of Intrapulmonary Percussive Ventilation (IPV) on Lung Compliance in Critically Ill Pediatric Patients Requiring Invasive Mechanical Ventilation.
Brief Title: IPV and Lung Compliance in Invasively Ventilated Children
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Steven and Alexandra Cohen Children's Medical Center (Individual)
Responsible Party: Sponsor
Other Study IDs: IRB# 24-0830
Record Dates: First submitted 2025-02-18; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome (PARDS); Pediatric Respiratory Diseases; Lung Compliance
Keywords: Lung Compliance; Pediatric; Pediatric Acute Respiratory Distress Syndrome (PARDS); Intrapulmonary Percussive Ventilation (IPV)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine if Intrapulmonary Percussive Ventilation (IPV) improves lung compliance in children receiving conventional invasive mechanical ventilation. The main questions it aims to answer are:

1. Does IPV improve lung compliance 15 minutes after and 3 hours after receiving one treatment in a heterogeneous group of pediatric patients?
2. Does IPV improve lung compliance in patients with Pediatric Acute Respiratory Distress Syndrome (PARDS), and what is the degree of change compared to those without PARDS?
3. What is the effect of IPV on lung compliance according to PARDS severity (mild-moderate disease vs. severe disease).
4. What is the incidence of adverse effects of IPV?

Participants will receive IPV because their medical team feels it will help their lung recovery and has already determined them to be safe candidates to receive this therapy, which is a standard airway clearance modality already routinely used in our PICU. Nothing additional will happen to participants as a result of this study. Enrolling in this study simply gives the study team permission to collect specific health information that identifies your child for research purposes, which may include results from medical tests found in their medical record and information from your child's bedside monitor and ventilator. This information will be collected before and after the IPV treatments to evaluate their response to the therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≤18 years old on conventional intermittent mandatory ventilation in the PICU that the physician deems is a candidate for IPV

Exclusion Criteria:

* The inability to accurately obtain ventilator measurements

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A heterogeneous population of pediatric patients <18 years old requiring conventional invasive mechanical ventilation and receiving IPV.
  We will also specifically identify and observe patients who meet criteria for Pediatric Acute Respiratory Distress Syndrome (PARDS) and compare the effects of IPV on lung compliance in this group relative to those without PARDS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic Compliance | Baseline (15 minutes before IPV treatment), 15 minutes after IPV treatment, and 3 hours after IPV treatment
  A measurement calculated and obtained from the patient's ventilator, averaged over 1 minute.

SECONDARY OUTCOMES:
Static Compliance (when applicable) | Baseline (15 minutes before IPV treatment), 15 minutes after IPV treatment, and 3 hours after IPV treatment
  A measurement calculated and obtained from the patient's ventilator using an inspiratory hold maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Sweberg, MD, Principal Investigator — Northwell Health
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No